CLINICAL TRIAL: NCT00133315
Title: TNFalfa Blocking Treatment of Spondylarthropathies - A Danish Multicenter Study of New Methods for Better Monitoring and Prognostifying Patients With Spondylarthropathies
Brief Title: TNFalfa Blocking Treatment of Spondylarthropathies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 232-001; KF 02-050/04
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2007-04-10 (Estimated); Status verified 2007-04

CONDITIONS: Spondylarthropathies; Ankylosing Spondylitis; Psoriatic Arthritis
MeSH Terms: conditions — Spondylarthropathies; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — Infliximab; Etanercept; Adalimumab

INTERVENTIONS:
Drug: Infliximab
Drug: Etanercept
Drug: Adalimumab

SUMMARY:
The purpose of the study is to establish a Danish cohort of spondylarthropathy (SpA) patients who are being treated with TNFalfa blockers. By following the TNFalfa blocking treated patients the researchers want to identify better biomarkers for disease activity and disease progression. In addition, the researchers want to identify predictors for disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Spondylarthropathies according to the European Spondylarthropathy Study Group (ESSG) criteria
* Sacroiliitis by X-ray or magnetic resonance imaging (MRI)
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)>3
* No signs of tuberculosis (TB)
* Sufficient contraception

Exclusion Criteria:

* Wish of pregnancy or nursing
* Previous treatment with TNFalfa blocker
* Disease-modifying anti-rheumatic drugs (DMARDs) other than methotrexate (MTX) later than 4 weeks before inclusion
* Steroid treatment later than 4 weeks before inclusion
* Immunosuppressing agents later than 4 weeks before inclusion
* Severe infections within 3 months
* HIV-infection
* Active hepatitis B and C
* Active or latent TB
* Severe chronic diseases
* Heart insufficiency (New York Heart Association [NYHA] 3 and 4)
* Malignancy
* Systemic lupus erythematosus (SLE) or SLE-like disease
* Abuse of narcotics or alcohol
* Major psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-09; Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inge Juul Soerensen, MD, Ph.D, Principal Investigator — Hvidovre University Hospital, Dept. of Rheumatology
Locations (9):
- Denmark (9):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Gentofte Municipality
  - Glostrup Hospital, Glostrup Municipality
  - Graasten Gighospital, Gråsten
  - Herlev Hospital, Herlev
  - Horsens Sygehus, Horsens
  - Hvidovre University Hospital, Hvidovre
  - Vejle Sygehus, Vejle

REFERENCES:
- [Derived] Pedersen SJ, Sorensen IJ, Lambert RG, Hermann KG, Garnero P, Johansen JS, Madsen OR, Hansen A, Hansen MS, Thamsborg G, Andersen LS, Majgaard O, Loft AG, Erlendsson J, Asmussen KH, Jurik AG, Moller J, Hasselquist M, Mikkelsen D, Ostergaard M. Radiographic progression is associated with resolution of systemic inflammation in patients with axial spondylarthritis treated with tumor necrosis factor alpha inhibitors: a study of radiographic progression, inflammation on magnetic resonance imaging, and circulating biomarkers of inflammation, angiogenesis, and cartilage and bone turnover. Arthritis Rheum. 2011 Dec;63(12):3789-800. doi: 10.1002/art.30627. PMID 22127697
- [Derived] Pedersen SJ, Sorensen IJ, Garnero P, Johansen JS, Madsen OR, Tvede N, Hansen MS, Thamsborg G, Andersen LS, Majgaard O, Loft AG, Erlendsson J, Asmussen K, Jurik AG, Moller J, Hasselquist M, Mikkelsen D, Skjodt T, Lambert R, Hansen A, Ostergaard M. ASDAS, BASDAI and different treatment responses and their relation to biomarkers of inflammation, cartilage and bone turnover in patients with axial spondyloarthritis treated with TNFalpha inhibitors. Ann Rheum Dis. 2011 Aug;70(8):1375-81. doi: 10.1136/ard.2010.138883. Epub 2011 May 8. PMID 21551511
- [Derived] Pedersen SJ, Sorensen IJ, Hermann KG, Madsen OR, Tvede N, Hansen MS, Thamsborg G, Andersen LS, Majgaard O, Loft AG, Erlendsson J, Asmussen K, Johansen JS, Jurik AG, Moller J, Hasselquist M, Mikkelsen D, Skjodt T, Hansen A, Ostergaard M. Responsiveness of the Ankylosing Spondylitis Disease Activity Score (ASDAS) and clinical and MRI measures of disease activity in a 1-year follow-up study of patients with axial spondyloarthritis treated with tumour necrosis factor alpha inhibitors. Ann Rheum Dis. 2010 Jun;69(6):1065-71. doi: 10.1136/ard.2009.111187. Epub 2009 Sep 9. PMID 19740906